CLINICAL TRIAL: NCT00590460
Title: Cd45 (Yth-24 and Yth 54) and Cd52 (Campath-1H) Monoclonal Antibody Conditioning Regimen for Allogeneic Donor Stem Cell Transplantation of Patients With Fanconi Anemia
Brief Title: Antibody Conditioning Regimen For Allogeneic Donor Stem Cell Transplantation Of Patients With Fanconi Anemia
Acronym: Mafia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Professor, Director Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-9938; NCT00058565 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Fanconi Anemia; Severe Aplastic Anemia
Keywords: Allogeneic Stem Cell Transplant; Fanconi Anemia; Severe Aplastic Anemia; fludarabine; campath; anti-CD45
MeSH Terms: conditions — Fanconi Anemia; Anemia, Aplastic | interventions — Alemtuzumab; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Study: Stem Cell Transplant (Experimental): CAMPATH-1H Anti-CD45 Fludarabine Stem Cell Infusion
  Interventions: Biological: CAMPATH-1H; Biological: Anti-CD45; Drug: Fludarabine; Procedure: Stem cell infusion

INTERVENTIONS:
Biological: CAMPATH-1H — Given intravenous on days -8, -7, and -6
  Other Names: Alemtuzumab
Biological: Anti-CD45 — Given intravenous on days -5, -4, -3 and -2
  dose is 400 micrograms/kg
Drug: Fludarabine — Given intravenous on days -8, -7, -6, -5 and -4
  Dose is 30 mg/m2
Procedure: Stem cell infusion — Stem cells are infused on day 0

SUMMARY:
The purpose of this study is to discover whether children and adults with Fanconi anemia (FA) can be safely and effectively transplanted with Human Leukocyte Antigen (HLA) mismatched (up to one haplotype), HLA-matched sibling, or unrelated donor stem cells, when leukocytolytic monoclonal antibodies are the sole conditioning agents (patients receiving an HLA mismatched transplant will receive Fludarabine as part of the conditioning regimen). Three monoclonal antibodies (MAb) will be used in combination. Two of them, YTH 24 and YTH 54 are rat antibodies directed against two contiguous epitopes on the CD45 (common leucocyte) antigen. They have been safely administered as part of the conditioning regimen for 12 patients receiving allografts (HLA matched and mismatched) at this center. They produce a transient depletion of >90% circulating leucocytes. The third MAb is Campath 1H, a humanized rat anti-CD52 MAb. This MAb has been widely used to treat B cell chronic lymphocytic leukemia (B-CLL) and more recently has been safely given at this and other centers as part of a sub-ablative conditioning regimen to patients with malignant disease. Because these MAb produce both profound immunosuppression and significant, though transient, myelodestruction we believe they may be useful as the sole conditioning regimen in patients with Fanconi anemia, in whom the use of conventional chemotherapeutic agents for conditioning produces a high rate of short and long term toxicity. We anticipate MAb mediated subablative conditioning will permit engraftment in a high percentage of these patients with little or no immediate or long term toxicity. Campath IH persists in vivo for several days after administration and so will be present over the transplant period to deplete donor T cells as partial graft versus host disease (GvHD) prophylaxis. Additional GvHD prophylaxis will be provided by administration of the medication FK506.

DETAILED DESCRIPTION:
If clinically feasible (no aplasia, no active malignancy), the recipients marrow will be harvested and cryopreserved as a back up for use if non-engraftment/rejection is followed by failure to undergo autologous reconstitution.

For HLA Mismatched donors, harvested peripheral blood stem cells will be enriched for CD34 cells using the Clinimacs CD34 Reagent system.

Fludarabine will be given as 5 daily intravenous infusions. Campath-1H will be given as 3 daily intravenous infusions and will be followed by Anti-CD45 which will be given as four daily intravenous infusions that will be completed two days prior to stem cell infusion. Diphenydramine will be administered intravenously every 4 hours during the period of the course of each infusion.

Day -8 Campath 1H as per CAGT SOP Fludarabine 30 mg/m2 -7 Campath 1H as per CAGT SOP Fludarabine 30 mg/m2 -6 Campath 1H as per CAGT SOP Fludarabine 30 mg/m2 -5 YTH 24/54 400ug/kg over 6 hr Fludarabine 30 mg/m2 -4 YTH 24/54 400ug/kg over 6 hr Fludarabine 30 mg/m2 -3 YTH 24/54 400ug/kg over 6 hr -2 YTH 24/54 400ug/kg over 6 hr -1 -0 Stem Cell Infusion

GVHD prophylaxis will be achieved through positive selection for CD34 resulting in > 3 log T cell depletion. Previous reports have indicated that there is a low frequency of severe (Grade II/IV) GvHD after haploidentical transplants if recipients receive stem cell populations containing <5 x 10e4 CD3 positive T cells. We hope to achieve such levels with our CD34 enrichment protocol. However, pharmacologic prophylaxis will be added if the CD34 selected product contains more than 5 x 10e4 CD3+ve T cells/kg recipient weight. In addition, Campath 1H persists in the recipient circulation through the immediate transplant period and will contribute anti-GVHD activity, in vivo.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Fanconi Anemia or other suspected DNA breakage/chromosomal instability syndromes, such as dyskeratosis congenita or Nijmegen breakage syndrome of all ages are eligible.

Diagnosis of Fanconi anemia confirmed by studies of peripheral blood or bone marrow sensitivity to mitomycin C or DEB or clinical evidence of other DNA breakage/chromosomal instability syndrome as determined by genetic testing or clinical diagnosis by a geneticist

Severe aplasia anemia as evidenced by a hypocellular bone marrow and at least 1 of the 3 criteria below: ANC < 500/mm3 Hemoglobin < 10 gm/dl with reticulocyte count < 1% Platelet count < 50,000/mm3

Availability of an HLA matched or mismatched (up to one haplotype) family member who has been documented not to have Fanconi anemia or of an unrelated HLA matched stem cell donor. Fully matched is defined at 6/6 match by high resolution DR based DNA typing.

Life expectancy greater than 6 weeks limited by diseases other than FA

Creatinine 2X normal for age or less

Karnofsky score 70% or more

Exclusion Criteria:

Patients with symptomatic cardiac disease, or evidence of significant cardiac disease by echocardiogram (i.e., shortening fraction less than 25%).

Patients with known allergy to rat serum products.

Patients with a severe infection that on evaluation by the Principal Investigator precludes ablative chemotherapy or successful transplantation.

Patients with severe personality disorder or mental illness.

Patients with documented HIV positivity.

Pregnant

NOTE: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator's discretion after approval by the CCGT Protocol Review Committee and the FDA Reviewer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2001-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Brenner, M.B., Ph.D.,, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Allo Stem Cell Transplant: Allogeneic Stem Cell Transplant
Period: Overall Study
Arm/Group | Allo Stem Cell Transplant
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group1: only one group
Arm/Group | Group1
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  <=5 years | 1
  Between 5 and 9 years | 2
  Between 10 and 15 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Donor Engraftment
Description: Number of patients with engraftment of at least 65% of donor cells 100 days after transplantation
Time Frame: 100 Days
Measure: Number; unit: participants
Groups:
- Allogeneic Stem Cell Transplant: Single Group: Allogeneic Stem Cell Transplant
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 5
participants | 2

2. Secondary Outcome: Number of Patients With Graft Failure
Description: Graft failure is defined as engraftment of less than 65% of donor cells 100 days after transplantation.
Time Frame: 100 days
Measure: Number; unit: participants
Groups:
- Allogeneic Stem Cell Transplant: Single Group - Allogeneic Stem Cell Transplant
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 5
participants | 3

3. Secondary Outcome: Patients With Treated Related Death
Description: Number of patients with treated related death
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Allo Stem Cell Transplant
Number analyzed (Participants) | 5
participants | 0

4. Secondary Outcome: Days to Absolute Neutrophil Count (ANC) of 500/mm3
Description: Number of days to Absolute neutrophil count (ANC) of 500/mm3
Time Frame: 30 Days
Measure: Median (Full Range); unit: days
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 5
days | 15 [14 to 16]

5. Secondary Outcome: Days to Platelet Count of 20,000/mm3 Without Transfusions
Description: Number of days to Platelet count of 20,000 / mm3 without transfusions
Time Frame: 30 Days
Population: Participants achieved a platelet count of 20,000 / mm3 without transfusions.
Measure: Median (Full Range); unit: days
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 2
days | 16 [14 to 18]

6. Secondary Outcome: Patients With Grade II - IV Acute Graft Versus Host Disease (GVHD)
Description: Number of patients with grade II - IV acute Graft versus Host Disease (GVHD)
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 5
participants | 0

7. Secondary Outcome: Number of Patients Alive at 1 Year Post Transplant
Description: Number of patients alive at 1 year post allogeneic stem cell transplant
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 5
participants | 5

8. Secondary Outcome: Patients With Limited Chronic GVHD From Day 100 to 365
Description: Number of patients with limited chronic GVHD from day 100 to 365
Time Frame: 365 days
Measure: Number; unit: participants
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 5
participants | 0

9. Secondary Outcome: Patients With Extensive Chronic GVHD From Day 100 to 365
Description: Number of patients with extensive chronic GVHD from day 100 to 365.
Time Frame: 365 days
Measure: Number; unit: participants
Groups:
- Allogeneic Stem Cell Transplant: only one group
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 5
participants | 0

10. Secondary Outcome: Patients With Grade III - IV Acute GVHD
Description: Number of patients with Grade III-IV acute GVHD
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group1
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group1 (N=5)
CNC hemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group1 (N=5)
Hypertension (Cardiac disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
AST (Hepatobiliary disorders) | 2 (4)
Picorna virus sinusitis (Infections and infestations) | 1 (1)
Herpes simplex type I (Infections and infestations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5)
Jaw Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes